CLINICAL TRIAL: NCT01218854
Title: A Comparison of Methods for Assisting Needle Angle Selection During Image-Guided Tissue Biopsy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 100217; 10-CC-0217
Record Dates: First submitted 2010-10-08; First posted 2010-10-11 (Estimated); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Lung Neoplasms; Liver Neoplasms; Kidney Neoplasms; Cancer
Keywords: Biopsy; Surgical Navigation; Image-guided Therapy; CT- Guided Biopsy; Cancer
MeSH Terms: conditions — Lung Neoplasms; Liver Neoplasms; Kidney Neoplasms; Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- B-NASS (Experimental): Block assisted needle angle selection system
  Interventions: Device: Needle angle measurement
- L-NASS (Experimental): laser assisted needle angle selection system
  Interventions: Device: Needle angle measurement
- MD-NASS (Experimental): mobile-device assisted needle angle selection system
  Interventions: Device: Needle angle measurement

INTERVENTIONS:
Device: Needle angle measurement — The tool for measuring the needle angles will be an FDA-approved EM tracking system. At no time will the needle enter tissue that it wouldn t have otherwise entered as neither system will be used to perform the biopsies at this time.

SUMMARY:
Background:

- Currently, standard procedures for biopsies that are guided by computed tomography (CT) imaging involve CT scans and a computer program to plan and illustrate where the physician will place the needle to obtain the required cells or tissue. Inserting the biopsy needle at the planned angle is not an easy task, because the appropriate angle of insertion must be estimated based on prior experience. Researchers are studying experimental techniques that might provide better guidance about the right angle to insert the biopsy needle and thereby improve the collection of the appropriate biopsy cells or tissue.

Objectives:

- To evaluate the effectiveness of two biopsy needle guidance methods in CT-guided tissue biopsy.

Eligibility:

- Individuals at least 18 years of age who are scheduled to have CT-guided tissue biopsy.

Design:

* Participants will have a tissue biopsy guided by CT scans and either a laser system or a plastic block to illustrate the appropriate angle of insertion. The skin will be numbed with anesthetic to minimize discomfort during the procedure.
* Before inserting the biopsy needle, the study physician will hold the needle in place so that a Food and Drug Administration-approved medical GPS (electromagnetic tracking) system can measure the needle angle as it enters the tissue.
* After the needle angle data has been collected, researchers will proceed with the actual biopsy procedure as it would normally occur, using standard methods.
* No additional treatment will be provided as part of this protocol.

DETAILED DESCRIPTION:
Background:

* Currently, standard/conventional CT-guided biopsies proceed as follows the physician:

  1. obtains a pre-procedural CT scan,
  2. plans the needle s angle based on this CT scan,
  3. selects the angle at which the needle should be inserted based on the pre-procedural CT scan,
  4. inserts the needle while aiming to replicate that planned needle angle by using only their visual-spatial abilities, and
  5. re-images the patient to confirm needle location followed by needle

     repositioning, if needed.
* Improving upon these standard methods of needle placement could have

widespread benefits (e.g. improved diagnostic tissue sampling, decreased

needle repositionings, etc.) We will be studying three needle angle selection systems. The laser-assisted needle angle selection system or LNASS, is a custom fabricated device that uses a Class II pointer similar to ones used for pointing at slides during lectures.

Objectives:

* To compare the angle difference between L-NASS (Method A) and the standard method (clinician intuition/conventional method)
* To compare the angle difference between B-NASS (Method B) and the standard method (clinician intuition)
* To compare the angle difference between the mobile device-NASS or MD-NASS (C) and the standard method (clinician intuition/conventional method)

Eligibility:

* Ages Eligible for Study: 18 Years and older
* Genders Eligible for Study: Both
* Inclusion:

  * Must be undergoing a scheduled CT-guided biopsy.
  * Must have ability to follow breathing instructions like holding breath (if procedure is to be performed without general anesthesia).
* Exclusion:
* No serious concurrent medical illness that would preclude the patient from making a rational informed decision on participation.
* Any known allergy to plastics or polymers (since the Ultem polymer could theoretically induce a rash in these patients, even though it is hypoallergenic).
* Pacemakers or automatic implantable cardiac defibrillators.
* Gross body weight above the CT table limit (450 pounds).

Design:

* Primary outcome measure for the first arm is:

  --The difference between planned and achieved needle angle of a laser-assisted needle angle selection system with the standard method (clinician s intuition or conventional method) of CT-guided biopsy.
* Primary outcome measure for the second arm is:

  --The difference between planned and achieved needle angle of a block with pre-drilled needle angles with the standard method (clinician s intuition or conventional method) of CT-guided biopsy
* Primary outcome for the third arm is:

  --The difference between planned and achieved needle angle of a mobile device-assisted needle angle selection system with the standard method (clinician's intuition or conventional method) of CT-guided biopsy.
* The tool for measuring the needle angles will be an FDA-approved electromagnetic tracking system, which tracks needle movement and position.
* These comparisons will be done as a bystander study.
* Needle guidance system will only be used initially to select the angle during a superficial, shallow needle insertion at the skin surface (less than 1 cm deep).
* At no time will the needle enter tissue that it wouldn t have otherwise entered as none of the system will be used to perform the biopsies at this time.
* The key portions of the procedure will not be altered in any substantive way.

ELIGIBILITY:
* INCLUSION CRITERIA:

Patients must fulfill all of the following criteria to be eligible for study admission:

* All patients must be undergoing a CT-guided biopsy.
* Age greater than 18 years.
* No serious concurrent medical illness that would preclude the patient from making a rational informed decision on participation.
* The ability to understand and willingness to sign a written informed consent form, and to comply with the protocol. If in question, an ethics consult will be obtained.
* Ability to follow breathing instructions like holding breath (if procedure is to be performed without general anesthesia).
* Patients must be actively enrolled on an NIH protocol and be scheduled for a CT-guided biopsy.

EXCLUSION CRITERIA:

* Patients with an altered mental status that precludes understanding or consenting for the biopsy procedure will be excluded from this study.
* Patients unlikely to be able to hold reasonably still on a procedure table for the length of the procedure.
* Patients with any known allergy to plastics or polymers (since the Ultem -polymer could theoretically induce a rash in these patients, even though it is hypoallergenic).
* Inability to follow breathing instructions, if without general anesthesia.
* Patients with pacemakers or automatic implantable cardiac defibrillators.
* Gross body weight above the CT table limit (450 pounds).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2012-03-20 (Actual); Primary Completion 2016-11-16 (Actual); Study Completion 2016-11-16 (Actual)

PRIMARY OUTCOMES:
Difference between L-NASS and standard method | Completion of study
  Data is currently undergoing analysis
Differnce between B-NASS and standard method | Completion of study
  Data is currently undergoing analysis
The difference between MD-NASS and standard method | Completion of study
  Data is currently undergoing analysis

CONTACTS AND LOCATIONS:
Overall Officials: Bradford J Wood, M.D., Principal Investigator — National Institutes of Health Clinical Center (CC)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided
It is not yet known if there will be a plan to make IPD available and still undecided.

REFERENCES:
- [Background] Miaux Y, Guermazi A, Gossot D, Bourrier P, Angoulvant D, Khairoune A, Turki C, Bouche E. Laser guidance system for CT-guided procedures. Radiology. 1995 Jan;194(1):282-4. doi: 10.1148/radiology.194.1.7997570.
- [Background] Pereles FS, Baker M, Baldwin R, Krupinski E, Unger EC. Accuracy of CT biopsy: laser guidance versus conventional freehand techniques. Acad Radiol. 1998 Nov;5(11):766-70. doi: 10.1016/s1076-6332(98)80260-2. PMID 9809074
- [Background] Jacobi V, Thalhammer A, Kirchner J. Value of a laser guidance system for CT interventions: a phantom study. Eur Radiol. 1999;9(1):137-40. doi: 10.1007/s003300050644. PMID 9933397
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2010-CC-0217.html